CLINICAL TRIAL: NCT03269500
Title: Evaluation of the Applicability of Personalized Tools About Nutrition Education for Malnourished Older People
Acronym: AlimAge
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2016/51
Record Dates: First submitted 2017-08-28; First posted 2017-08-31 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Malnutrition of Mild Degree

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- malnourished older people: The hospitalized elderly with swallowing and/or Mastication problems.
  Interventions: Other: use of nutrition education tools

INTERVENTIONS:
Other: use of nutrition education tools — Use of different nutrition education tools :
  * General advice: feeding seniors
  * Oral supplementation: instructions for use
  * Information about enriched food
  * Food modified in texture: chopped masticatory disorders, chopped swallowing disorders, co-mingled
  * How should I drink? : With stimulus, texture syrup / nectar, velvety texture, texture compote / cream
  * Recipe booklets for people to easily eat (chewing disorders) or recipe with molded texture (swallowing disorders)

SUMMARY:
Describe the frequency of use of nutrition education tools for undernourished older people

DETAILED DESCRIPTION:
The description of the population will identify the characteristics of patients who use the tools and guide their use in patient care. To realize an impact assessment, It necessary to identify specific criteria for inclusion. It is important initially to assess the use of the nutritional tools. The assessment of performance (obstacles and understanding), will be used to improve tools to optimize their use.

ELIGIBILITY:
Inclusion Criteria:

* Subject of 75 years or more.
* Hospitalized geriatric day hospital.
* Living at home, within a radius of 40 km around the hospital Xavier Arnozan.
* Subject or caregiver (s) read, understand and speak the french.
* Undernutrition (criteria of the French high authority for health (HAS) 2007)
* Agreed to participate in the study: compendium of the opposition

Exclusion Criteria:

* Subject not wishing to participate in the study,
* MMSE (Mini Mental State Examination) < 20, without presence of a caregiver with no cognitive problems scoring.
* Identified palliative care.
* Presenting a contraindication to oral feeding.
* Presence of supply of enteral or parenteral.
* Presence with a diagnosis of severe psychiatric pathology.
* Already participating in a study on undernutrition.
* One against medical advice.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: malnourished elderly present on hospital day care
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2018-08-07 (Actual); Study Completion 2018-08-07 (Actual)

PRIMARY OUTCOMES:
Frequency of use of the booklet and platelets | Day 14
  number of use per week

SECONDARY OUTCOMES:
Evaluation of the knowledge following the delivery of the tools | Day 14
  Number of response "Yes" for 24 items about the tools
Instrumental Activities of Daily Living | Day 1
  Score of Instrumental Activities of Daily Living
Assessment of quality of life scale | Day 1
  Score of EQ-5D

CONTACTS AND LOCATIONS:
Overall Officials: Ornella SARRY, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Bordeaux University Hospital, Pessac, France

IPD SHARING:
Plan to Share IPD: No